CLINICAL TRIAL: NCT03841565
Title: Phase II Trial of Daratumumab Retreatment in Patients With Relapsed Multiple Myeloma
Brief Title: Daratumumab, Pomalidomide, and Dexamethasone in Treating Patients With Relapsed Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: There are no patients enrolled on this study and all efforts are being discontinued.
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-MY-1601; NCI-2019-00386 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-MY-1601 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2021-08

CONDITIONS: Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pomalidomide, daratumumab, dexamethasone) (Experimental): Patients receive pomalidomide PO QD on days 1-21 and daratumumab IV on days 1, 8, 15, and 22 of cycles 1-2, days 1-15 of cycles 3-6, and day 1 of subsequent cycles. Patients also receive dexamethasone PO on days 1, 8, 15, and 22 of cycles 1-12. Cycles every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Daratumumab; Drug: Dexamethasone; Drug: Pomalidomide

INTERVENTIONS:
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase II trial studies how well daratumumab, pomalidomide, and dexamethasone work in treating patients with multiple myeloma that has come back (relapsed). Immunotherapy with daratumumab may induce changes in body's immune system and may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as pomalidomide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving daratumumab with dexamethasone and pomalidomide may work bettering in treating patient compared to dexamethasone and pomalidomide alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (partial response [PR], very good partial response [VGPR], complete response [CR], or stringent complete response [sCR]) of daratumumab retreatment in combination with pomalidomide and dexamethasone (DPd) in patients with relapsed refractory multiple myeloma.

SECONDARY OBJECTIVES:

I. To assess progression free survival and overall survival associated with retreatment with daratumumab in combination with pomalidomide and dexamethasone (DPd) in patients with relapsed and refractory multiple myeloma.

II. To determine the toxicities associated with retreatment with daratumumab in combination with pomalidomide and dexamethasone (DPd).

OUTLINE:

Patients receive pomalidomide orally (PO) once daily (QD) on days 1-21 and daratumumab intravenously (IV) on days 1, 8, 15, and 22 of cycles 1-2, days 1-15 of cycles 3-6, and day 1 of subsequent cycles. Patients also receive dexamethasone PO on days 1, 8, 15, and 22 of cycles 1-12. Cycles every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for every 3 months until subsequent treatment or progressive disease, then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Calculated creatinine clearance (using Cockcroft-Gault equation) >= 30 mL/min (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 14 days prior to registration)
* Untransfused platelet count >= 75,000/mm^3 (obtained =< 14 days prior to registration)
* Hemoglobin >= 8.0 g/dL (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (except for patients with Gilbert's syndrome) (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (obtained =< 14 days prior to registration)
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Bone marrow >= 30% plasma cells
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Relapsed multiple myeloma (MM) requiring treatment who have previously received a daratumumab alone or in a daratumumab containing combination and

  * Had at least a partial response to therapy, and had disease progression on or within 60 days of discontinuation
  * At least 3 months should have elapsed since last exposure to daratumumab
  * Patients must have been previously exposed to both a proteasome inhibitor and an immunomodulatory imide drug (IMiD)

    * Examples of proteasome inhibitors:

      * Bortezomib, carfilzomib, ixazomib, marizomib, oprozomib
    * Examples of IMiD's:

      * Thalidomide, lenalidomide, pomalidomide
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to follow strict birth control measures

  * Female patients: If they are of childbearing potential, agree to one of the following:

    * Practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
  * Male patients: even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

    * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
    * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Willing to follow the requirements of the Pomalyst Risk Evaluation and Mitigation Strategy (REMS) program
* Willing to provide bone marrow and blood samples for planned research

Exclusion Criteria:

* Refractory to pomalidomide
* Concurrent amyloid light chain (AL) amyloidosis with organ involvement
* Diagnosed or treated for another malignancy =< 2 years prior to registration or previously diagnosed with another malignancy and have any evidence of residual disease. NOTE: Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Any of the following because this study involves an investigational agent, whose genotoxic, mutagenic and teratogenic effects, on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other concurrent chemotherapy, or any ancillary therapy considered investigational. NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Major surgery =< 14 days prior to registration
* Evidence of current uncontrolled cardiovascular conditions, including hypertension, cardiac arrhythmias, congestive heart failure, unstable angina, or myocardial infarction =< 6 months. Note: Prior to entry, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Known human immunodeficiency virus (HIV) positive
* Known hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Seropositive for human immunodeficiency virus (HIV)

  * Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
  * Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts or investigator's brochure) or known sensitivity to mammalian-derived products
* Known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal
* Known moderate or severe persistent asthma within the past 2 years or currently has uncontrolled asthma of any classification
* Total bilirubin =< 1.5 x ULN (except for patients with Gilbert's syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Best overall response rate to the therapy | Up to 3 years
  A success will be defined as a partial response or better noted as the objective status on two consecutive evaluations. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Overall survival time | From registration to death due to any cause, assessed up to 3 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Progression-free survival | From registration to the earliest date of documentation of disease progression on initial therapy or death due to any cause, assessed up to 3 years
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Incidence of adverse events | Up to 3 years
  Will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

OTHER OUTCOMES:
Proportion of minimal residual disease (MRD) negativity | Up to 3 years
  MRD will be assessed on bone marrow aspirate in all patients achieving complete response (CR) or stringent CR (sCR). The proportion of patients who achieve MRD negative status will be estimated by the number of patients who are MRD negative divided by the total number of evaluable patients who achieve CR or sCR. Exact binomial 95% confidence intervals for the true MRD negative rate will be calculated.
Changes in clonal population and CD38 expression | Baseline up to 3 years
  Will be summarized descriptively by median, min, max, and interquartile range at each time point. Changes from baseline to after treatment will be assess using paired analyses, including Wilcoxon signed rank tests.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K Kumar, Principal Investigator — Academic and Community Cancer Research United
Locations (5):
- United States (5):
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - State University of New York Upstate Medical University, Syracuse, New York
  - McLeod Regional Medical Center, Florence, South Carolina